CLINICAL TRIAL: NCT04107831
Title: Physical Function in Patients With Chronic Obstructive Pulmonary Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: Norwegian Fund for Postgraduate Training in Physiotherapy (Other); Western Norway University of Applied Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HaukelandUH- 2019/852
Record Dates: First submitted 2019-09-15; First posted 2019-09-27 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2023-03

CONDITIONS: COPD
Keywords: Pulmonary rehabilitation; Exercise; Field walk test; Physical performance test
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary rehabilitation (Experimental): Participants who are participating in a 6-week pulmonary rehabilitation program are enrolled in the study.
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — Pre-post test design

SUMMARY:
The aims of the study are to examine the responsiveness of, and the correlation between field walk tests and physical performance test in patients with chronic obstructive pulmonary disease (COPD) after participating in pulmonary rehabilitation.

DETAILED DESCRIPTION:
Patients with COPD who are participating at pulmonary rehabilitation (PR) at Haukeland University Hospital will be asked and consecutive enrolled to the study. Before and after PR the six-minute walk test, incremental- and endurance shuttle walk test, 30 sec sit-to-stand test and stair test will be used to evaluate change in physical capacity and -performance.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with COPD, Forced expiratory volume in 1 sec (FEV1)/Forced vital capacity (FVC) <0.7 and FEV1<80% of predicted value.
* Able to walk corridor and stairs
* Norwegian speaking

Exclusion Criteria:

* COPD exacerbations requiring medical treatment last 4 weeks prior to inclusion led to deferment of inclusion
* Not safe to exercise (e.g unstable angina)
* mental illness and drug abuse that makes group treatment not suitable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-09 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test | up to 6 weeks
  Change from baseline to 6 weeks in 6 minute walk distance in meter is primary outcome

SECONDARY OUTCOMES:
Incremental Shuttle walk test | up to 6 weeks
  Change from baseline to 6 weeks in walk distance in meter is the outcome
Endurance shuttle walk test | up to 6 weeks
  Change from baseline to 6 weeks in time in second is the outcome
30 second sit to stand test | up to 6 weeks
  Change from baseline to in number of repetition is the outcome
Stair test | Up to 6 weeks
  Change from baseline to 6 weeks in time of the test is the outcome: 18 steps are walked up and down three times as fast as possible. Time in sec. is measured.

CONTACTS AND LOCATIONS:
Overall Officials: Else Sterndorff, Director, Study Director — Haukeland University Hospital, Dept. of Physiotherapy
Locations (1):
- Bente Frisk, Sandsli, Norway

IPD SHARING:
Plan to Share IPD: Undecided